CLINICAL TRIAL: NCT03100721
Title: Pain Neuroscience Education as a Complement to Physiotherapy in Patients With Chronic Musculoskeletal Pain: a Non-randomized Controlled Trial
Brief Title: Pain Neuroscience Education in Chronic Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Collaborators: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Principal Investigator, Alejandro Luque-Suarez, PhD, University of Malaga
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNE in MSK
Record Dates: First submitted 2017-03-22; First posted 2017-04-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: Education; Chronic pain; Musculoskeletal pain; Self-efficacy
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNE+Physiotherapy (Experimental): Pain neuroscience education (PNE) can be defined as an educational session or sessions describing the neurobiology and neurophysiology of pain, and pain processing by the nervous system. It will be applied one time (at baseline). Physiotherapy includes kinesitherapy and exercises.
  Interventions: Behavioral: PNE+Physiotherapy
- Physiotherapy (Active Comparator): Physiotherapy includes kinesitherapy and exercises.
  Interventions: Procedure: Physiotherapy

INTERVENTIONS:
Behavioral: PNE+Physiotherapy — Physiotherapy cover kinesitherapy and exercises techniques. Besides that it will be covered the understanding and acknowledgement about how pain is processed.
  Arms: PNE+Physiotherapy
Procedure: Physiotherapy — Physiotherapy cover kinesitherapy and exercises techniques.
  Arms: Physiotherapy

SUMMARY:
Chronic musculoskeletal pain (CMP) is highly prevalent, disabling and with high socio-economic costs, with many negative effects on quality of life. CMP affects the ability to perform work, social, recreational and domestic tasks by changing the mood and concentration of this population that suffers.

In a study carried out in 2010, 17% of the Spanish population had experienced pain in the last month and according to the severity of symptoms 12% felt severe , 64% moderate and 24% mild pain. In this same study it is specified that 61% was due to back pain, 29% due to neck pain and 23% due to shoulder pain.

Pain neuroscience education (PNE) has been shown as an effective treatment strategy in increasing knowledge and understanding of neurobiology, neurophysiology and pain processing, modifying beliefs about it, improving patient skills and encouraging to the accomplishment of physical and social activities in different chronic pathologies.

DETAILED DESCRIPTION:
Study design and setting: The design of the present study will be a quasi-experimental study with 2 follow-ups (one month and four months after intervention) that will be performed between Apr 2018 and Apr 2020 in public health system in Malaga, Spain. The outcomes will be assessed at baseline (t0), one month (t1) and four months after the physiotherapy treatment begins (t2). Written informed consent will be acquired for all participants prior to their participation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* Chronic Musculoskeletal Pain according to the ACCTION-APS Pain Taxonomy (AAPT), included chronic axial musculoskeletal low back pain

Exclusion Criteria:

* Chronic postoperative musculoskeletal pain and chronic musculoskeletal pain related to a traumatic injury six months before the beginning of the trial
* Inability to provide written informed consent and/or complete questionnaires in Spanish.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline self-efficacy at 1 and 4 months | 1 and 4 months
  This outcome will be measured with the Chronic Pain Self-Efficacy Scale

SECONDARY OUTCOMES:
Change from Baseline pain and pain interference at 1 and 4 months | 1 and 4 months
  This outcome will be measured with the Graded Chronic Pain Scale
Change from Baseline analgesic medication at 1 and 4 months | 1 and 4 months
  This outcome will be measured checking digital medical history

OTHER OUTCOMES:
Change from Baseline pain knowledge at 1 and 4 months | 1 and 4 months
  This outcome will be measured with the revised Neurophysiology of Pain Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Luque Suarez, PhD, Principal Investigator — University of Malaga
Locations (1):
- UGC Las Lagunas, Mijas Costa, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No